CLINICAL TRIAL: NCT06787911
Title: The Efficacy and Safety of Donafenib Combined With Anti-PD-1 Antibody for Neoadjuvant Therapy in Locally Advanced Thyroid Cancer: a Phase II Study
Brief Title: Donafenib Combined With Anti-PD-1 Antibody for Neoadjuvant Therapy in Locally Advanced Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yu Wang (Other)
Responsible Party: Sponsor-Investigator, Yu Wang, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPM-DTC
Record Dates: First submitted 2024-11-30; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Patients receive Donafenib and PD-1 antibody Sintilimab
  Interventions: Drug: Donafeib with Sintilimab

INTERVENTIONS:
Drug: Donafeib with Sintilimab — Patients receive Donafenib and PD-1 antibody Sintilimab

SUMMARY:
This study is a single-arm intervention study. Locally advanced differentiated thyroid carcinoma patients receive neoadjuvant therapy with Donafenib and PD-1 antibody Sintilimab and those who can undergo surgery after neoadjuvant therapy receive surgical treatment. The aim of the study is to evaluate the efficacy and safety of Donafenib combined with PD-1 antibody in neoadjuvant therapy of locally advanced thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily enroll and sign a written informed consent form;
2. Age>=18 years old,<=80 years old, regardless of gender;
3. Locally advanced differentiated thyroid carcinoma (DTC) diagnosed by pathological histology;
4. Locally advanced DTC is defined as meeting at least one of the criteria: surgery is expected to be difficult to complete R0/R1 resection; AJCC defined T4 stage: any size of tumor infiltrating beyond the thyroid capsule to the subcutaneous soft tissue, throat, trachea, esophagus, recurrent laryngeal nerve, tumor invades the prevertebral fascia or surrounds the carotid or mediastinal vessels.
5. Voluntarily undergo tumor biopsy/operation at enrollment and exit.
6. Have not received any anti-tumor treatment in the past;
7. According to the evaluation criteria for the efficacy of solid tumors (RECIST version 1.1), there should be at least one imaging measurable lesion. Lesions located within the radiation field of previous radiotherapy can be considered measurable if confirmed to have progressed;
8. The physical condition (PS) score of the Eastern Cancer Collaborative Group (ECOG) is 0-2 points;
9. Expected survival time>3 months;
10. Female patients with fertility (referring to those who have not undergone menopause or surgical sterilization) must have a negative serum pregnancy test result within 7 days before the study drug administration;
11. Female or male patients with fertility must take reliable contraceptive measures during the study drug use period and within 60 days after the last medication use;
12. Normal function of major organs, i.e. meeting the following criteria: Blood routine examination (no blood transfusion or G-CSF used within 14 days prior to screening): a) Hemoglobin>=90 g/L; b) Absolute neutrophil count (ANC)>=1.5 × 109/L; c) Platelet count>=80 × 109/L; Blood biochemistry test (no albumin used within 14 days prior to screening): d) Total bilirubin<=1.5 x Upper limit of normal value (ULN); e) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)<=2.5 x ULN (ALT or AST<=5 x ULN allowed for subjects with liver metastasis); f) Creatinine<=1.5 x ULN; Coagulation function: g) International standardized ratio (INR) or prothrombin time (PT)<=1.5 x ULN; h) Activated partial thromboplastin time (APTT)<=1.5 x ULN; Others: i) Urinary protein<2+(if urinary protein>=2+, 24-hour urine protein quantification can be performed, and 24-hour urine protein quantification<1.0g can be included in the group).j)Myocardial enzyme profiles were within the normal range (simple laboratory abnormalities not clinically significant were also allowed to be included)

Exclusion Criteria:

1. Other histological subtypes of thyroid cancer (such as undifferentiated carcinoma, myeloid carcinoma, lymphoma, or sarcoma) that are not associated with DTC;
2. Patients who undergo thyroid cancer radical surgery again;
3. Central nervous system metastasis and/or cancerous meningitis with clinical symptoms, and a history of leptomeningeal carcinoma;
4. Within the first 5 years of randomization, cancer with a different primary site or histological type from thyroid cancer, or cancer coexisting with thyroid cancer but with a different primary site or histological type, except for cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (non-invasive tumors, carcinoma in situ, and tumor invasion of the lamina propria);
5. Previous or current congenital or acquired immunodeficiency disease;
6. Active or previously documented autoimmune disease or inflammatory disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, Hypophysitis, hyperthyroidism or hypothyroidism, asthma requiring bronchodilator treatment, etc.), patients with vitiligo or asthma that has been completely resolved in childhood, without any intervention in adulthood can be included;
7. Have a history of severe mental illness in the past;
8. Suffering from diseases that affect the absorption, distribution, metabolism, or clearance of investigational drugs (such as severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorders, etc.); Previous or concomitant medication/treatment:
9. Has undergone major surgery (as defined by the researcher) within 4 weeks prior to enrollment, or is expected to require major surgery during the study treatment period;
10. Have received iodine-131 ablation or other local anti-tumor treatments within the past 3 months, or plan to undergo systemic anti-tumor treatment or external irradiation or other interventional treatments during the medication period of this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or have used mitomycin C within 6 weeks before receiving the investigational drug treatment). The use of levothyroxine for TSH inhibition and thyroid hormone supplementation therapy is not prohibited;
11. Previously received organ or allogenic bone marrow transplantation;
12. Previously received targeted therapy drugs targeting VEGF, including but not limited to anlotinib, apatinib, bevacizumab, etc;
13. Previously received immune therapy drugs including but not limited to anti CTLA-4, anti PD-1, anti PD-L1, anti PD-L2, anti CD137. Therapeutic anti-tumor vaccines are not included;
14. Systemic immunosuppressive drug treatment has been used within 2 weeks before enrollment, or systemic immunosuppressive drug treatment is expected to be required during the study period, except for the following cases:

    1. Intranasal, inhaled, topical or local injection (such as intra-articular injection) corticosteroids;
    2. The dose does not exceed 10 mg/day of prednisone or other equivalent systemic corticosteroids;
    3. Prophylactic use of corticosteroids for hypersensitivity reactions;
15. Simultaneously taking drugs that may prolong QTc and/or induce apical torsion transition ventricular tachycardia (Tdp) or affect drug metabolism;

    Security:
16. The patient has a known or suspected history of allergies to donafinib or similar drugs, or a history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or allergies to excipients of the study drug;
17. Imaging shows that the tumor has invaded important blood vessels, or the investigator determines that the patient's tumor is highly likely to invade important blood vessels during treatment and cause fatal bleeding;
18. Active bleeding or abnormal coagulation function, with a tendency to bleed or undergoing thrombolysis, anticoagulation, or antiplatelet therapy;
19. Have a history of gastrointestinal bleeding within the past 4 weeks or have a clear tendency for gastrointestinal bleeding (such as known local active ulcer lesions, fecal occult blood++, if continuous fecal occult blood++, gastroscopy should be performed), or other conditions determined by the researcher that may cause gastrointestinal bleeding (such as severe gastric fundus/esophageal varices);
20. Have experienced gastrointestinal perforation, abdominal fistula, or abdominal abscess within the past 6 months;
21. Have experienced thrombosis or thromboembolic events within the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc;
22. Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting surgery within the past 6 months, congestive heart failure (New York Heart Association NYHA grade>2), poorly controlled or requiring pacemaker treatment for arrhythmia, and uncontrolled hypertension (systolic blood pressure>=140 mmHg and/or diastolic blood pressure>=90 mmHg);
23. Active infections, including: a) AIDS virus (HIV/2 antibody) positive; b) Active hepatitis B (HBsAg positive and abnormal liver function); c) Active hepatitis C (HCV antibody positive or HCV RNA ≥ 103 copies/ml with abnormal liver function); d) Active tuberculosis; e) Other uncontrollable active infections (CTCAE V5.0>level 2);
24. Other significant clinical and laboratory abnormalities, which the researchers believe affect the safety evaluation, such as uncontrollable diabetes, chronic kidney disease, peripheral neuropathy of grade II or above (CTCAE V5.0), thyroid dysfunction, etc;
25. Has not yet recovered from surgery, such as the presence of unhealed incisions or serious postoperative complications;
26. Within 4 weeks prior to enrollment or possibly during the study period, receive any attenuated live vaccines;
27. Pregnant or lactating women, as well as female or male patients with fertility who are unwilling or unable to take effective contraceptive measures;

    Other:
28. Have a history of alcohol, psychotropic drugs, or other substance abuse within the past 6 months;
29. Have received clinical trials of other drugs or medical devices within 4 weeks prior to enrollment. TSH inhibition therapy is not prohibited;
30. Unable to follow the research protocol for treatment or follow up on schedule;
31. Any other researcher deemed ineligible for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From enrollment to the end of treatment at 4 weeks
  The proportion of patients with complete response (CR) and partial response (PR) to the total number of evaluable cases.

SECONDARY OUTCOMES:
R0/R1 resection rate | From enrollment to the end of treatment at 4 weeks
  The rate of patients who receive R0 or R1 resection surgery after neoadjuvant treatment in all patients undergo surgery.
Progression free survival | 5 years after surgery
  The time from surgery to tumor progression, including local-regional recurrence and distant metastasis
Tumor recurrence time | 5 years after surgery
  Time from treatment to the first date received CR or PR status
disease control rate | 5 years after surgery
  The percentage of patients who received CR、PR or SD status of all patients enrolled
3-year local recurrence-free survival | From enrollment to the end of treatment at 3 years
  3-year local recurrence-free survival
5-year local recurrence-free survival | From enrollment to the end of treatment at 5 years
  5-year local recurrence-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided